CLINICAL TRIAL: NCT03094481
Title: Comparison of Interscalene vs. Superficial Cervical Block vs. Combination of Both Blocks for Analgesia After Operative Repair of Midshaft and Lateral Clavicle Fractures
Brief Title: Interscalene vs. Superficial Cervical Block vs. Combination for Analgesia After Clavicle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul McHardy, Assistant Professor, Staff Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 036-2016
Record Dates: First submitted 2017-03-15; First posted 2017-03-29 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Clavicle Fracture
MeSH Terms: interventions — small cardioactive peptide B; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be blinded except for the specific anesthesiologist performing the nerve blocks. This person will not be involved in providing further care (administering anesthesia) nor data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- US guided SCPB medial fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5% (1:200,000) epinephrine. 10ml injected for ultrasound guided Superficial Cervical Plexus Block at C4 or C5.
  Interventions: Procedure: SCPB; Drug: Bupivacaine hydrogen chloride , epinephrine
- US guided ISB medial fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5%(1:200,000) epinephrine. 10ml injected for ultrasound guided Interscalene Brachial Plexus Block at C5 or C6.
  Interventions: Procedure: ISB; Drug: Bupivacaine hydrogen chloride , epinephrine
- US guided SCPB + ISB medial fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5% (1:200,000) epinephrine. 10ml injected for ultrasound guided Superficial Cervical Plexus Block at C4 or C5. 10ml injected for ultrasound guided Interscalene Brachial Plexus Block at C5 or C6.
  Interventions: Procedure: SCPB + ISB; Drug: Bupivacaine hydrogen chloride , epinephrine
- US guided SCPB lateral fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5% (1:200,000) epinephrine. 10ml injected for ultrasound guided Superficial Cervical Plexus Block at C4 or C5.
  Interventions: Procedure: SCPB; Drug: Bupivacaine hydrogen chloride , epinephrine
- US guided ISB lateral fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5%(1:200,000) epinephrine. 10ml injected for ultrasound guided Interscalene Brachial Plexus Block at C5 or C6.
  Interventions: Procedure: ISB; Drug: Bupivacaine hydrogen chloride , epinephrine
- US guided SCPB + ISB lateral fracture (Active Comparator): Bupivacaine hydrogen chloride Inj 0.5% (1:200,000) epinephrine. 10ml injected for ultrasound guided Superficial Cervical Plexus Block at C4 or C5. 10ml injected for ultrasound guided Interscalene Brachial Plexus Block at C5 or C6.
  Interventions: Procedure: SCPB + ISB; Drug: Bupivacaine hydrogen chloride , epinephrine

INTERVENTIONS:
Procedure: SCPB — Bupivacaine hydrogen chloride Inj 0.5% epinephrine. 10ml injected for US guided Superficial Cervical Plexus Block at C4 or C5.
  Other Names: Superficial Cervical Plexus
  Arms: US guided SCPB lateral fracture; US guided SCPB medial fracture
Procedure: ISB — Bupivacaine hydrogen chloride Inj 0.5% epinephrine. 10ml injected for US guided Interscalene Brachial Plexus Block at C5 or C6.
  Other Names: Interscalene Brachial Plexus
  Arms: US guided ISB lateral fracture; US guided ISB medial fracture
Procedure: SCPB + ISB — Bupivacaine hydrogen chloride Inj 0.5% epinephrine. 10ml injected for US guided SCPB at C4 or C5 + 10ml injected for ISB at C5 or C6.
  Other Names: Superficial Cervical Plexus & Interscalene Brachial Plexus
  Arms: US guided SCPB + ISB lateral fracture; US guided SCPB + ISB medial fracture
Drug: Bupivacaine hydrogen chloride , epinephrine — Bupivacaine hydrogen chloride Inj 0.5% (1:200,000) epinephrine

SUMMARY:
The optimal analgesic peripheral nerve block (or combinations thereof) are undefined for clavicle fractures, the most frequent fracture in the human population. This goal of this study is to determine whether interscalene block (ISB), superficial cervical plexus block (SCPB), or both provide the best analgesia for lateral and midshaft clavicular fractures, respectively.

DETAILED DESCRIPTION:
Clavicle fractures are relatively common injuries that occur most often in young active males and elderly individuals. They are often a result of direct trauma to the shoulder, typically from a fall. Clavicle fractures represent 5-10% of all fractures and represent the most frequent fracture in the human population. Midshaft fractures account for 69-85% of the clavicle fractures, distal shaft fractures 12-28%. (1) Analgesia for clavicle fractures can be challenging for anaesthetists secondary to the complex and varied innervation in this region. Literature describing the innervation of the clavicle and overlying skin is heterogeneous with the C3 to C6 nerve roots being involved. The clavicle itself has been reported to be innervated either by C4 or by C5 and C6 (subclavian nerve) nerve roots. (2) Regional anaesthesia for intraoperative and postoperative analgesia of clavicle fractures employs several possible, commonly used approaches. The contemporary literature surrounding the optimal regional anaesthetic technique for clavicle surgery which can provide superior postoperative analgesia and minimize systemic agents intraoperatively is lacking Currently there are only small case series or case reports published. Peripheral nerve blocks used to anesthetize the clavicle include SCPB, ISB, and combined SCPB-ISB. Larger, systematic trials have not yet been performed to our knowledge and as recently as one year ago a call for more evidence in this area of regional anaesthesia was published in the American Society of Regional Anesthesia and Pain Medicine. The purpose of this study is to compare analgesic outcomes after the common regional anesthetic techniques (ISB versus SCPB versus both).

ELIGIBILITY:
Inclusion Criteria:

* undergoing open reduction and internal fixation of clavicle fracture (midshaft or lateral)

Exclusion Criteria:

* lack of patient consent
* contra-indication to upper extremity peripheral nerve block (eg. severe pulmonary dysfunction)
* inability to lie supine for nerve block
* polytrauma
* pre-existing neurologic deficit in operative upper extremity
* allergy to amide local anesthetic
* contralateral phrenic nerve dysfunction
* chronic opioid use (>30mg daily oral morphine equivalent)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10-21 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain measurement using NRS in PACU | 1 hour post-op
  Numeric Rating Scale for Pain upon discharge from Post-anesthetic Care Unit

SECONDARY OUTCOMES:
Pain measurement using NRS at Discharge | 4 hours post-op
  Numeric Rating Scale for Pain upon discharge from hospital
Opioid consumption in morphine equivalence | 4 hours post-op
  Total postoperative opioid consumption from end of operation to hospital discharge
Satisfaction using rating scale | 4 hours post-op
  Patient satisfaction with postoperative analgesia at time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Paul McHardy, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faldini C, Nanni M, Leonetti D, Acri F, Galante C, Luciani D, Giannini S. Nonoperative treatment of closed displaced midshaft clavicle fractures. J Orthop Traumatol. 2010 Dec;11(4):229-36. doi: 10.1007/s10195-010-0113-z. Epub 2010 Oct 9. PMID 20936323
- [Background] Choi DS, Atchabahian A, Brown AR. Cervical plexus block provides postoperative analgesia after clavicle surgery. Anesth Analg. 2005 May;100(5):1542-1543. doi: 10.1213/01.ANE.0000149049.08815.00. No abstract available. PMID 15845732
- [Background] Tran DQ, Tiyaprasertkul W, Gonzalez AP. Analgesia for clavicular fracture and surgery: a call for evidence. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):539-43. doi: 10.1097/AAP.0000000000000012. PMID 24121609